CLINICAL TRIAL: NCT06989385
Title: CORALINE - Correlation Between Physiological and Clinical Variables and Failure of Non-Invasive Respiratory Support in Patients With Acute Respiratory Failure
Acronym: CORALINE
Status: Recruiting | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Roberto Tonelli, Assistant Professor, University of Modena and Reggio Emilia
Other Study IDs: UModenaReggio2025
Record Dates: First submitted 2025-04-24; First posted 2025-05-25 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Failure
Keywords: Acute respiratory failure; High flow nasal cannula; Non-invasive ventilation; Inspiratory effort
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is an observational study. Interventions are standard of care and include: High-flow nasal oxygen (HFNO) Non-invasive ventilation (NIV) Pnose monitoring — No experimental interventions are administered as part of the study.

SUMMARY:
This observational study aims to evaluate the relationship between clinical and physiological variables and the failure of non-invasive respiratory support (NIRS), including high-flow nasal oxygen (HFNO) and non-invasive ventilation (NIV), in patients with acute respiratory failure (ARF), both hypoxemic and/or hypercapnic. The study includes both retrospective and prospective components. Retrospective data will be collected from patient charts, while prospective data will be collected at defined time points during clinical care. The primary outcome is NIRS failure, defined as the need for orotracheal intubation. Secondary outcomes include in-hospital and 90-day mortality, ICU and hospital length of stay, and duration of non-invasive and invasive support.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalization in the Respiratory Medicine Unit at AOU Policlinico di Modena
* Acute respiratory failure (hypoxemic and/or hypercapnic) with PaO₂/FiO₂ < 300 mmHg
* Undergoing treatment with HFNO or NIV

Exclusion Criteria:

* Immediate need for invasive ventilation upon admission
* Known neuromuscular disease
* Pregnancy
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Respiratory Disease Unit of the University of Modena and Reggio Emilia
Sampling Method: Non-Probability Sample
Enrollment: 325 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of failure of non-invasive respiratory support | 30 days
  Number of patients experiencing NIRS failure (defined as escalation to another NIRS modality, need for orotracheal intubation, or death) over the total number of patients.

SECONDARY OUTCOMES:
Clinical impact | From enrollment to 90 days
  Mortality

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Policlinico di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided